CLINICAL TRIAL: NCT06957249
Title: Clinical Study to Evaluate the Tooth Whitening Efficacy of a Colgate Toothpaste With 5% Hydrogen Peroxide and Fluoride Compared to a Toothpaste With 0% Hydrogen Peroxide and Fluoride Over a One-Week Period.
Brief Title: Clinical Study to Evaluate the Tooth Whitening Efficacy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2025-04-WHT-5OW-FL-BGS
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-05

CONDITIONS: Whitening
Keywords: hydrogen peroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test 1 Toothpaste (Experimental): fluoride toothpaste
  Interventions: Drug: Optic White 5%HP ActivShine Toothpaste
- Test 2 Toothpaste (Active Comparator): fluoride toothpaste
  Interventions: Drug: Crest3DWhite Advanced Radiant Mint Toothpaste

INTERVENTIONS:
Drug: Optic White 5%HP ActivShine Toothpaste — 0.76% MFP toothpaste
  Arms: Test 1 Toothpaste
Drug: Crest3DWhite Advanced Radiant Mint Toothpaste — 0.243% NaF toothpaste
  Arms: Test 2 Toothpaste

SUMMARY:
Optic White 5%HP ActivShine TP vs Crest3D White TP (head-to-head whitening clinical) The objective of this study is to evaluate the tooth whitening efficacy of a Colgate toothpaste with 5% Hydrogen Peroxide and Fluoride compared to a toothpaste with 0% Hydrogen Peroxide and Fluoride over a one-week period.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form;
* Male and female subjects 18-70 years old, inclusive;
* Good general health and good oral health based on the opinion of the study investigator;
* All maxillary natural permanent anterior teeth (6-11) must be present;
* Availability for the duration of the study;
* Minimum average Vita Extended Bleachedguide 3D-Master shade score of 17 ≥ or darker.

Exclusion Criteria:

* Presence of orthodontic appliances and/or any anterior tooth with a prosthetic crown, veneer, or deemed non-vital;
* Obvious signs of periodontal disease, rampant caries, or any condition that the dental examiner considers exclusionary from the study;
* Five or more carious lesions requiring immediate care;
* Concurrent participation in another clinical study;
* Self-reported pregnant and/or lactating women;
* History of allergies or sensitivity to tooth whitening products, hydrogen peroxide, personal care consumer products, or their ingredients;
* Restorations on the teeth to be scored which may interfere with scoring procedures;
* Have used a professional whitening product within one (1) year and/or had a dental prophylaxis (professional dental cleaning) within thirty (30) days prior to the start of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-05-03 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Tooth color measurement | baseline, day 1, day 3, day 7
  Changes in Tooth color determined by examiner use of Vita Extended Bleachedguide 3D-Master® (29 tabs)

CONTACTS AND LOCATIONS:
Overall Officials: John Gallob, DMD, Principal Investigator — Consumer Research Consulting, LLC
Locations (1):
- Consumer Research Consulting, LLC, Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: No